CLINICAL TRIAL: NCT05809739
Title: FLASH Study: Effectiveness and Safety of STYLAGE® HYDRO in the Treatment of Face, Neckline Area and Neck
Brief Title: Effectiveness and Safety of STYLAGE® HYDRO in the Treatment of Face, Neckline Area and Neck
Acronym: FLASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIV-STYL-HYD-01; 21E3942 (Other: Dermscan)
Record Dates: First submitted 2023-02-17; First posted 2023-04-12 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Aging
Keywords: hyaluronic acid; Injection; Healthy subjects; Prospective; Single arm; ISR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Device: STYLAGE® Hydro
  1 mL up to 2.0 mL per area will be injected in the face, neckline and neck (optionally) at each injection session.
  Interventions: Device: STYLAGE Hydro

INTERVENTIONS:
Device: STYLAGE Hydro — 3 sessions of injections (J0, J14 and J28)

SUMMARY:
FLASH Study is a Post-Market Follow-Up PCMF designed to evaluate the tolerance and efficacy of STYLAGE Hydro by using a satisfaction questionnaire.

DETAILED DESCRIPTION:
This is a prospective, in open, single arm and multicentric study designed to evaluate the tolerance and efficacy of STYLAGE Hydro.

Patients will be injected up to 2 mL of STYLAGE Hydro per area at each session. Three injection sessions 2 weeks apart are planned: one at visit 1 (D0), one at visit 2 (W2) and one at visit 3 (W4).

Proportions of subjects who are satisfied on the face 6 weeks after treatment initiation will be assessed. For each question of the questionnaire, the subjects who are satisfied are defined as subjects who rated "Somewhat agree", "Agree" or "Totally agree". Global aesthetic improvement according to independent evaluator and subjects' satisfaction will also be done during other visits. Safety parameters will be evaluated during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject.
2. Sex: female.
3. Age: between 30 and 70 years.
4. Subject having given freely and expressly her informed consent and data privacy consent.
5. Subject with signs of cutaneous dryness and lack of elasticity on the face, on the neckline area and if applicable on the neck (if neck is planned to be treated) following investigator assessment.
6. Subject willing to have photographs of the face, neck and neckline taken.
7. Subject psychologically able to understand the study related information and to give a written informed consent.
8. Subject affiliated to a health social security system.
9. Subject agreeing not to receive another aesthetic procedure (e.g., laser, dermabrasion, surgery, deep chemical peeling, surface peel, tensor threads, injection with a filling product) on the face, the neckline area and if applicable on the neck (if neck is planned to be treated) during the whole study.
10. Female of childbearing potential should use a medically accepted contraceptive regimen since at least 12 weeks before screening visit and during the whole study.
11. Subject agreeing to keep their usual cleansing / care products during the whole study period.
12. Subject agreeing to apply a SPF50 cream during non-intensive exposure to sunlight.

Exclusion Criteria:

1. Pregnant or breastfeeding woman or planning a pregnancy during the study.
2. Subject with a tattoo, a scar, moles, too many hairs or anything on the studied zones which might interfere with the evaluation.
3. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
4. Subject in a social or sanitary establishment.
5. Subject participating to another research on human beings or who is in an exclusion period of one.
6. Subject having received 6000 euros indemnities for participation in researches involving human beings in the 12 previous months, including participation in the present study. (France only)
7. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results.
8. Subject suffering from autoimmune disease and/or immune deficiency.
9. Subject suffering from inflammatory and/or infectious cutaneous disorders in or near the studied zones (herpes, acne, mycosis, papilloma…). Subject with recurrent herpes is eligible if asymptomatic at time of inclusion.
10. Subject having history of hypersensitivity to hyaluronic acid or to one of the components of the tested device, anaesthetic product or antiseptic solution.
11. Subject having history of anaphylactic shock or severe and/or evolutive / unstable / recent allergy.
12. Subject with a past history of streptococcal disease, such as acute rheumatic fever or recurrent sore throats.
13. Subject predisposed to develop keloids or hypertrophic scars.
14. Subject prone to develop inflammatory skin conditions or having tendency to bleeding disorders.
15. Subject having received treatment with a laser on the face, the neckline area or if applicable the neck within the past 6 months prior to screening visit.
16. Subject having received a superficial, medium, or deep peeling on the face, the neckline area or if applicable the neck within the past month, 3 or 12 months respectively prior to screening visit.
17. Subject having received injection with a reticulated hyaluronic acid (HA), on the face, the neckline area or if applicable the neck within the past 12 months prior to screening visit.
18. Subject having received injection with a non-reticulated hyaluronic acid (HA) or botulinum toxin on the face, the neckline area or if applicable the neck within the past 6 months prior to screening visit.
19. Subject having received at any time injection with a slowly resorbable filling product (polylactic acid, calcium hydroxyapatite, combinations of HA and hypromellose, HA and dextran microbeads or HA and TriCalcium Phosphate (TCP), …),a non-resorbable filling product (polyacrylamide, silicone, combination of methacrylic polymers and collagen, polymer particles, …) or tensor threads on the face, the neckline area or if applicable the neck.
20. Subject having started or changed her oral contraceptive or any other hormonal treatment during 12 weeks prior to screening visit.
21. Subject using medication such as aspirin, NSAIDs (ibuprofen, ketoprofen, naproxen…), platelet aggregation inhibitors, anticoagulants, vitamin C within one week prior to injection visit (V1) and agreeing not to take such treatments within 1 week prior to the second (V2) and third injections (V3).
22. Subject having history of immunosuppressors taking.
23. Subject undergoing a topical treatment on the test area or a systemic treatment:

    * Anti-histamines during the 3 days prior to injection visit (V1) and agreeing not to take such treatment during the study as far as possible;
    * Corticoids during the 4 weeks prior to screening visit;
    * Retinoids during the 6 months prior to screening visit.
24. Subject having changed her topical cleansing / care products within the month prior to screening visit.
25. Intensive exposure to sunlight or UV-rays within the previous month and foreseen during the study.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Subject's satisfaction with STYLAGE® HYDRO on the face | 6 weeks after treatment initiation
  Proportions of subjects who are satisfied after treatment using a questionnaire (question 1 to 7)

SECONDARY OUTCOMES:
Subject's satisfaction with STYLAGE® HYDRO on the face | 6, 9 and 12 weeks after treatment initiation
  Proportions of subjects who are satisfied after treatment using a questionnaire (since question 8 on week 7) and mean changes from baseline in subject's scores for satisfaction using the FACE-Q satisfaction with skin questionnaire.
  For FACE-Q questionnaire, the minimum score of 1 means a worse outcome and the maximum score of 4 means a better outcome.
Subject's satisfaction with STYLAGE® HYDRO on the neckline area and if applicable on the neck | 6, 9 and 12 weeks after treatment initiation
  Proportions of subjects who are satisfied on the neckline area and if applicable on the neck after treatment using a questionnaire
Investigator's satisfaction on the face, the neckline area and if applicable on the neck | 6 and12 weeks after treatment initiation
  Proportions of subjects for whom the investigator is satisfied on the face, the neckline area and if applicable on the neck after treatment using a questionnaire
Effectiveness of STYLAGE® HYDRO in improving the subject's aesthetic appearance on the face, the neckline area and if applicable the neck | 6, 9 and 12 weeks after treatment initiation for subject and at 7 and 12 weeks after treatment initiation for investigator
  Proportions of GAIS responders on the face, the neckline area and if applicable on the neck as assessed by subject and investigator
Effectiveness of STYLAGE® HYDRO on skin thickness on the face and neckline area | 6 and 12 weeks after treatment initiation
  Mean change from baseline in average thickness of the epidermis and dermis (mm) on the face and neckline area after treatment using DermaScan C USB®
Effectiveness of STYLAGE® HYDRO on skin density on the face and neckline area | 6 and 12 weeks after treatment initiation
  Mean changes from baseline in proportion of non-echogenic tissues (%) on the face and neckline area after treatment using DermaScan C USB®
Mean change in average roughness on the face | 6 and 12 weeks after treatment initiation
  Mean change from baseline in average roughness (micrometer) on the face after treatment using Dermatop®
Mean change in average height of the roughness on the face | 6 and 12 weeks after treatment initiation
  Mean change from baseline in average height of the roughness (micrometer) on the face after treatment using Dermatop®
Mean change in maximum height of the roughness profile on the face | 6 and 12 weeks after treatment initiation
  Mean change from baseline in maximum height of the roughness profile (micrometer) on the face after treatment using Dermatop®
Mean change in arithmetic mean height of the roughness on the face and neckline area | 6 and 12 weeks after treatment initiation
  Mean change from baseline in arithmetic mean height (micrometer) on the face and neckline area after treatment using C-Cube®
Mean change in root mean square height of roughness on the face and neckline area | 6 and 12 weeks after treatment initiation
  Mean change from baseline in root mean square height (dimensionless) on the face and neckline area after treatment using C-Cube®
Mean change in ratio of the developed interfacial area on the face and neckline area | 6 and 12 weeks after treatment initiation
  Mean changes from baseline in ratio of the developed interfacial area (%) on the face and neckline area after treatment using C-Cube®
Mean change in the depth of crow's feet wrinkles | 6 and 12 weeks after treatment initiation
  Mean changes from baseline in the severity of crow's feet wrinkles after treatment using Dermatop®
Injection pain with STYLAGE® HYDRO | Day 0, Day 14 and Day 28
  Mean pain scores during injection assessed by subject on a 100 mm Visual Analogue Scale (VAS).
  Minimum value is 0 mm and maximum value is 100 mm. Higher scores mean a worse outcome.
Incidence of injection site reactions and adverse events | Through study completion, an average of 14 weeks
  Product tolerance will be assessed by collection of Injection Site Reactions (ISRs) after each injection session and of Adverse Events (AEs) throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Zunaid M. ALLI, MD, Principal Investigator — Harley Street Hospital
Locations (2):
- France (2):
  - Eurofins Dermscan, Aix-en-Provence
  - Eurofins Dermscan Pharmascan, Villeurbanne

IPD SHARING:
Plan to Share IPD: No